CLINICAL TRIAL: NCT04472130
Title: Biomarkers in Neurodegenerative Diseases
Brief Title: Neurodegenerative Diseases Registry
Acronym: NDD Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vincent Mok (Other)
Responsible Party: Sponsor-Investigator, Vincent Mok, Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: CRE-2019.371
Record Dates: First submitted 2020-06-25; First posted 2020-07-15 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Neurodegenerative Diseases; Parkinson Disease; Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: Neurodegenerative Diseases; Parkinson Disease
MeSH Terms: conditions — Neurodegenerative Diseases; Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Plasma, blood cells, cerebrospinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Early idiopathic Parkinson's Disease: 200 patients with iPD based on Movement Disorder Society clinical diagnostic criteria for Parkinson's disease with disease onset less than 5 years
- Non-early idiopathic Parkinson's Disease: 200 patients with iPD based on Movement Disorder Society clinical diagnostic criteria for Parkinson's disease with disease onset more than 5 years
- Multiple System Atrophy: 100 patients with Multiple System Atrophy based on Second consensus statement on the diagnosis of MSA
- Progressive Supranuclear Palsy: 100 patients with Progressive Supranuclear Palsy based on Clinical research criteria for diagnosis of PSP
- Alzheimer's Disease: 100 patients with Alzheimer's Disease by Diagnostic and Statistical Manual of Mental disorder, Fifth edition (DSM-5) criteria
- Motor Neuron Disease: 200 patients with Motor Neuron Diseases by revised El Escorial criteria or Awaji ALS criteria
- Small Vessel Disease: 200 patients with cerebral Small Vessel Diseases
- Frontotemporal Dementia: 100 patients with Frontotemporal Dementia by International consensus criteria for behavioral variant FTD (FTDC) or Primary Progressive Aphasia by Gorno-Tempini
- Healthy Control: 200 age and sex matched healthy controls

SUMMARY:
With the increase in life expectancy of our population due to advancement of medical diagnosis and treatments, the incidence of age dependent neurodegenerative diseases increased, including Alzheimer's disease (AD), parkinsonian syndromes (PS), small vessel disease (SVD) and motor neuron disease (MND). In spite of the progress of knowing the pathogenesis of various neurodegenerative diseases at molecular and genetic level, they are still very incompletely understood and often cause diagnostic and therapeutic challenges to physicians. Due to the overlapping presentation and similar brain pathology, especially in the early stage of the diseases, it is difficult to differentiate idiopathic Parkinson's disease (iPD) from atypical parkinsonian syndromes, such as multiple system atrophy (MSA) and progressive supranuclear palsy (PSP). Similarly, distinguishing AD from other dementia syndromes including frontotemporal dementia (FTD), dementia with Lewy Bodies (DLB), corticobasal degeneration (CBD) and vascular dementia can be difficult. It is necessary to develop accurate and comprehensive diagnostic tests to properly prognosticate the diseases, start treatments in early stage of the diseases and maximize the accuracy of drug trials for more effective preventive and therapeutic measures for these neurodegenerative diseases.

Therefore, the registry aims to generate a large database of cognitive, behavioral, lifestyle and psychological information of the subjects who suffered from neurodegenerative diseases, as well as to examine the genetic basis of neurodegenerative diseases to help decode the pathogenic mechanisms of the diseases. The registry may provide important information to understand symptom development of the neurodegenerative diseases, in which may help physicians to diagnose the diseases more accurately and provide better treatment plans.

DETAILED DESCRIPTION:
This is a cohort study. It involves baseline, 1st follow up visit and 2nd follow up visit. At baseline visit, all participants will go through a list of assessments and questionnaires and blood taking. Follow-up visit(s) will be scheduled every one to two years, in which the same set of assessments and questionnaires will be administered.

1. Clinical assessments and questionnaires

   Different clinical assessments would be administered depending on the group that the participant belongs to:
   * Hoehn and Yahr Stage and the Unified Parkinson's Disease Rating Scale (UPDRS) for iPD, PSP and SVD patients with parkinsonism features
   * Unified MSA Rating Scale (UMSARS) for MSA
   * Levodopa Equivalent Dosage for medication burden for parkinsonian syndromes patients
   * Amyotrophic lateral sclerosis functional rating scale revised (ALSFRS-R), body weight and forced vital capacity (FVC) for MND group
   * Montreal Cognitive Assessment Hong Kong version (HK-MoCA), Olfactory Identification Test (OIT) and Farnsworth-Munsell 100 Hue test for all groups

   Video taking would be administered to record participants' eye movement if necessary. For example, video of eye movement is useful to rate MSA patients' ocular motor dysfunction, such as gaze-evoke nystagmus.

   Patients with parkinsonian syndromes will fill in a set of questionnaires, including demographic information, medical history, history and current medications, wearing-off questionnaire, impulsiveness questionnaire, Buss-Perry Aggression Questionnaire (BPAQ), rapid eye movement sleep behavior disorder questionnaire (RBDQ), Epworth Sleepiness Scale (ESS), Morningness-Eveningness Questionnaire (MEQ), Insomnia Severity Index (ISI), Beck's Scale for Suicide Ideation (BSSI), Scales for Outcomes in Parkinson's Disease-Autonomic questionnaire (SCOPA-AUT), Hospital Anxiety and Depression Scale (HADS), Patient Health Questionnaire (PHQ9), lifestyle and life history, and occupation history.
2. Blood sampling Blood taking would be carried out at Prince of Wales Hospital and will be processed and transported to the laboratory according to standard procedure.

   Venous blood samples are collected into 6 EDTA tubes and 1 Heparin tube. The volume of total blood samples will not exceed 23ml. Serum is obtained within 1 hour by centrifugation at 3,000 rpm for 10 min and stored at -70°C until laboratory evaluation for proteomics, SERS and other biochemical and genetics studies.
3. Sub-studies Selected participants in the cohort groups, especially those with early disease onset and/or familial cases, would proceed to sub-studies which include brain MRI, brain PET, lumbar puncture and/or skin biopsy. Subjects are voluntary to join one or more sub-studies.

ELIGIBILITY:
Inclusion Criteria:

* Age should be between 18-80 years old.

Exclusion Criteria:

* Patients with ongoing central nervous system infection and/or acute stroke or active brain tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited in neurology outpatient clinic in Prince of Wales Hospital, Hong Kong, who meet the inclusion and exclusion criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
the score change in Unified Parkinson's Disease Rating Scale (UPDRS) | baseline visit, 2 years after baseline visit, 4 years after baseline visit
  The Unified Parkinson's Disease Rating Scale (UPDRS) would be administered to assess disease severity for iPD, PSP and SVD patients with parkinsonism features
the score change in Unified MSA Rating Scale (UMSARS) | baseline visit, 2 years after baseline visit, 4 years after baseline visit
  The Unified MSA Rating Scale (UMSARS) would be administered to assess disease severity for patients with MSA
the score change in Montreal Cognitive Assessment Hong Kong version (HK-MoCA) | baseline visit, 2 years after baseline visit, 4 years after baseline visit
  Montreal Cognitive Assessment Hong Kong version (HK-MoCA) is used to assess participants' cognitive functions for all groups

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mok, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong